CLINICAL TRIAL: NCT00282061
Title: Synchronization and Desynchronization Between Circadian Rhythms in Patients With Delayed Sleep Phase Syndrome (DSPS)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: SHEBA-04-3497-YD-CTIL
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2006-12-15 (Estimated); Status verified 2006-01

CONDITIONS: Delayed Sleep Phase Syndrome
Keywords: 3 conditions in a within-subject design:; 1-ad-lib sleep wake; 2-forced morning wake-up; 3- ad-lib sleep wake after treatment with melatonin
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Melatonin

INTERVENTIONS:
Drug: Melatonin

SUMMARY:
This study's first aim is to widen the knowledge of the characteristics of delayed sleep phase disorder (DSPS) by focusing on the circadian rhythms of appetite regulation factors and their phase relations to the cycles of sleep-wake, melatonin, cortisol and body temperature. This study's second aim is to assess the influence of forced morning awakening, as a daily struggle faced by DSPS patients, upon the synchronization of these variables in DSPS patients. The investigators hypothesize that the chronic incompatibility between the endogenous sleep-wake rhythm of the DSPS patients and the morning wakefulness, as a social demand, may impair the synchronization between the different rhythms, as findings indicate in normal subjects under jet lag. And finally, the third aim of the study is to assess the influence of successful treatment with melatonin upon the phase locations of circadian rhythms of studied measures and the synchronization between them. These measures will be assessed in a controlled study, for 36 hours (sampled every 2 hours) under three distinct experimental conditions: first, under free sleep-wake conditions (ad-libitum bedtime and arousal); second, under restricted sleep-wake conditions (enforced morning wake-up); and finally, after 12 weeks of melatonin treatment.

DETAILED DESCRIPTION:
Method:

Subjects:

A total of 20 subjects, 10 diagnosed as DSPS patients and 10 matched healthy controls with a proven normal sleep-wake cycle.

Exclusion criteria for the recruitment would be body mass index (BMI) higher than 28 or lower than 22, shift-work, or chronic disease and chronic medication use.

Procedure:

Experiment 1- A comparison between 10 normal rhythm and 10 DSPS subjects under restricted sleep-wake schedule

Stage 1: 10 day actigraphic monitoring under restricted sleep schedule (using alarm clocks): DSPS patients will be awakened at 7:00 a.m., and control subjects will be awakened at 3:00 a.m.

Stage 2: A 36 hour monitoring of the following measures: body temperature, melatonin, cortisol, Ghrelin, subjective hunger sensation and eating behavior. The subjects will be provided with ad-libitum food and will be instructed to eat whatever they like, whenever they feel hungry.

Experiment 2- A comparison between 10 normal rhythm and 10 DSPS subjects under ad-libitum sleep conditions

Stage 1: A 10 day actigraphic monitoring under ad-libitum sleep schedule. Patients will be instructed to go to sleep whenever they feel tired and avoid any means of unnatural awakening.

Stage 2: similar to experiment 1.

Experiment 3- Examination of DSPS patients under melatonin administration and ad libitum sleep, after 12 weeks of treatment

Stage 1: A 10 day actigraphic monitoring under ad-libitum sleep schedule. Patients will be instructed to go to sleep whenever they feel tired and avoid any means of unnatural awakening. Melatonin will be taken according to the medical instruction (usually at 22:00).

Stage 2: similar to experiment 1.

Measurements:

Subjective hunger sensation will be measured with Visual Analogue Scale ratings for appetite assessment (Flint et al. 2000; Oh et al. 2002; Parker et al. 2004).

Timing of meals and eating behavior will be recorded by the experimenter during the 36-hr monitoring.

Sleep-wake rhythm (normal or DSPS) will be determined using the Actiwatch wrist activity monitoring system (Actiwatch, Cambridge Neurotechnology LTD.)

Plasma levels of Ghrelin: will be sampled every 2 hours for 36 hours. An intravenous catheter will be placed on the subject's arm 30 minutes prior to the first blood sampling. Blood samples will be collected with chilled Vacutainer EDTA tubes and immediately centrifuged. Plasma Ghrelin will be measured using commercial radioimmunoassay (RIA- Phoenix Pharmaceuticals).

Salivary levels of Melatonin and Cortisol: Saliva will be collected by placing wool swab of plain Salivettes (Sarstedt, Disposable Products, Regency Park, Adelaide) into the mouths of the subjects with chewing for 5 min. Saliva samples will be taken at a total of 18 time points over a 36-h period for each subject. The samples will be kept in Salivette tubes in the refrigerator at ±4 ºC until the end of each 24-h period. The Salivette tubes will be centrifuged for 15 min at 3000 ´g and the samples frozen at -20 ºC until assayed.

Melatonin treatment: Subjects with DSPS in the treatment group will be treated with melatonin according to a standard protocol for 3 months before the experiment.

Oral temperature: will be measured using standard medical mercury thermometer, placed under the tongue for 3 minutes at a total of 18 time points over a 36-h period right after the saliva sample collection.

Analysis Assays of Melatonin and cortisol: Melatonin in saliva was measured by a direct radioimmunoassay (RIA). The kit is manufactured by LDN GmbH & Co, KG, Nordhorn Germany (Cat-No: DSL-BA-1200) and is specially made for the quantitative determination of melatonin in saliva. The cross-reactivity of the assay for N-acetylserotonin, 5-methoxytryptophol, and 5-methoxytryptamine is 0.80%, 0.70%, and 0.08%. Serotonin, 5-methoxyindole-3-acetic acid is < 0.01%, respectively. The sensitivity of the assay is 1 ng/L. The intra- and inter-variations are 11.3% and 12%, respectively. Salivary cortisol concentrations were measured with a competitive solid-stage radioimmunoassay [Coat-A-Count, Diagnostic Products Corp (DPC)]. The protocol followed the instructions of Coat-Count Free Cortisol in Saliva kit from DPC.

Ghrelin assay: Plasma immunoreactive ghrelin levels will be measured in duplicate using a commercial radioimmunoassay (RIA) that uses 125I-labeled bioactive ghrelin as a tracer and a rabbit polyclonal antibody raised against full-length octanoylated human ghrelin (Phoenix Pharmaceuticals, Belmont, CA).

Setting:

The experiments will take place at the Institute for Sleep and Fatigue medicine, the Chaim Sheba Medical Center, Tel Hashomer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of DSPS

Exclusion Criteria:

* BMI higher than 28 or lower than 22
* Shift-work
* Chronic disease and chronic medication use

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Dagan, MD, PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- The Institute for Sleep and Fatigue Medicine, Sheba Medical Center, Tel Litwinsky, Israel